CLINICAL TRIAL: NCT00643604
Title: Rapid Switch From Intravenous Epoprostenol to Intravenous Remodulin® (Treprostinil Sodium) in Patients With Stable Pulmonary Arterial Hypertension in the Outpatient Clinic: Safety, Efficacy and Treatment Satisfaction
Brief Title: Rapid Switch From Flolan to Remodulin in the Outpatient Clinic
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to availability of eligible subjects at center and enrollment competition with other studies.
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIV-PH-413
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Results first posted 2013-06-21 (Estimated); Last update posted 2024-01-03 (Actual); Status verified 2013-06

CONDITIONS: Hypertension, Pulmonary
Keywords: Pulmonary arterial hypertension; treatment satisfaction; rapid switch; remodulin; Quality of life
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — treprostinil; Epoprostenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treprostinil sodium (Experimental): all subjects had switched from IV epoprostenol to IV treprostinil sodium
  Interventions: Drug: treprostinil sodium

INTERVENTIONS:
Drug: treprostinil sodium — rapid switch from intravenous epoprostenol on CADD ambulatory pump to intravenous treprostinil sodium
  Other Names: Remodulin; Flolan

SUMMARY:
The purpose of this 8-week study is to compare the effects of switching from therapy with epoprostenol or Flolan to IV Remodulin. This study will also assess the effect that changing to Remodulin will have on patient satisfaction with their treatment and impact on quality of life.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH), which is defined as an elevation in pulmonary arterial pressure and pulmonary vascular resistance, is a severe hemodynamic abnormality common to a variety of diseases and syndromes. Elevation in pulmonary arterial pressure causes an increase in right ventricular afterload, impairing right ventricular function and ultimately leading to inactivity and death. The goal of PAH treatment is to lengthen survival time, to ameliorate symptoms of PAH and to improve health related quality of life (HRQOL).

Remodulin® (treprostinil sodium), a stable analogue of prostacyclin, possesses potent pulmonary and systemic vasodilatory and platelet anti-aggregatory actions in vitro and in vivo. Recently, Remodulin received FDA approval for intravenous therapy based upon bioequivalence of the IV and SC routes of administration. Remodulin is more chemically stable than epoprostenol and may offer potential safety and convenience advantages compared to intravenous epoprostenol that may impact Health Related Quality of Life (HRQOL) and/or patient satisfaction. Unlike epoprostenol, Remodulin does not need to be mixed daily and is stable at room temperature eliminating the need for ice packs. Furthermore, since Remodulin remains in the body longer than epoprostenol (4 hrs instead of less than 5 minutes) there is less risk of cardiovascular collapse from a sudden interruption of infusion, such as a line clog. In an open-label study in Europe, patients who were using a type of portable medication pump called the CADD Legacy pump were rapidly switched from Flolan to Remodulin with no serious side effects. This study will examine effects of switching from therapy with epoprostenol or Flolan to IV Remodulin and compare changes in HRQOL and treatment satisfaction before and after rapid switch from epoprostenol to Remodulin in patients with pulmonary hypertension using the CADD legacy pump.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 years and 70 years of age
* Be male or if female, be physiologically incapable of childbearing or practicing an acceptable method of birth control (women of childbearing potential must have a negative pregnancy test).
* Have a current World Health Organization (WHO) functional classification of II-III status
* Diagnosis of one of the following WHO Classifications of pulmonary hypertension: Group 1 pulmonary arterial hypertension (IPAH, FPAH, APAH);Group 3 pulmonary hypertension associated with lung disease (Mild interstitial lung disease associated with predominant features of right heart failure as seen in Group 1 PAH patients); Group 4 pulmonary hypertension due to chronic thromboembolic pulmonary hypertension (CTEPH)
* In the opinion of the investigator, be hemodynamically stable with no signs or symptoms of disease progression
* Be receiving intravenous epoprostenol therapy for at least three months and a stable dose for at least one month prior to Baseline.
* Have a central intravenous catheter in place.
* Have a baseline six-minute walk distance of at least 150 meters.
* Be optimally treated with conventional pulmonary hypertension therapy and clinically stable for at least one month prior to baseline assessments.
* Be mentally and physically capable of learning to administer Remodulin using an intravenous infusion pump.

Exclusion Criteria:

* Be a nursing or pregnant woman
* Have had a new type of chronic therapy (including but not limited to oxygen, a different category of vasodilator, a diuretic, digoxin, bosentan, sildenafil) for pulmonary hypertension added within the last month.
* Have any PAH medication discontinued within the week prior to study entry.
* Received any prostacyclin or prostacyclin analog except epoprostenol in the past 3 months.
* Have an on-going central venous line infection within the past 30 days.
* Have evidence of predominant left-sided heart disease
* Have any other disease that is associated with pulmonary hypertension (e.g. sickle cell anemia, schistosomiasis).
* Have a musculoskeletal disorder (e.g. arthritis, artificial leg, etc.) or any other disease, which is thought to limit ambulation, or be connected to a machine, which is not portable.
* Have uncontrolled systemic hypertension as evidenced by a systolic blood pressure greater than 160 mmHg or diastolic blood pressure greater than 100 mmHg.
* Be receiving an investigational drug, have in place an investigational device, or have participated in an investigational drug study within the past 30 days.
* Have the presence of any physiological or psychological condition that contraindicates the administration of Remodulin.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2008-03; Primary Completion 2010-01 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victor Tapson, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled in March 2008. Given the limited availability of eligible subjects at the investigative center (stable PH patients on stable epoprostenol therapy) and competition for enrollment by other studies, after an extended recruitment period during which no new subjects were enrolled, the study was subsequently closed.
Groups:
- Treprostinil Sodium: treprostinil sodium : all subjects underwent a rapid switch from intravenous epoprostenol on CADD ambulatory pump to intravenous treprostinil sodium
Period: Overall Study
Arm/Group | Treprostinil Sodium
Started | 7
Completed | 6
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 43.6 (32-58) [32 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 7
Pulmonary Arterial Hypertension (PAH) etiology [Number; unit: participants]
  Idiopathic PAH | 5
  Collagen Vascular Disease | 1
  Portal Hypertension | 1
World Health Organization (WHO) functional Class at time of transition [Number; unit: participants] — Class I: No limitation of physical activity. Class II: Slight limitation of physical activity. Class III: Marked limitation of physical activity. Class IV: Inability to carry out any physical activity without symptoms.
  participants
    Class II | 5
    Class III | 2
Baseline 6 Minute Walk Distance (6MWD) [Mean (Full Range); unit: meters] | 466.6 [343 to 565]

OUTCOME MEASURES:

1. Primary Outcome: Change in Six Minute Walk Distance
Time Frame: Baseline and Week 8
Population: Two subjects had a Week 8 visit that was outside of the visit window and are included in the summary. One subject died prior to Week 8 assessments.
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 6
meter | -14 (63.7)
Statistical Analysis 1: Comparison: Treprostinil Sodium; Changes between Baseline and Week 8 were assessed using the Wilcoxon signed rank test. A two-sided p value of < 0.05 was considered statistically significant. No imputation was used for missing values; Test type: Superiority or Other; p = 0.69, Wilcoxon signed-rank test

2. Secondary Outcome: Change in WHO Functional Classification
Description: Class I: No limitation of physical activity. Class II: Slight limitation of physical activity. Class III: Marked limitation of physical activity. Class IV: Inability to carry out any physical activity without symptoms.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 6
participants
  Improved | 0
  No change | 5
  Worsened | 1
Statistical Analysis 1: Comparison: Treprostinil Sodium; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 1.00, Wilcoxon signed-rank test

3. Secondary Outcome: Change in Borg Dyspnea Score Immediately After Six Minute Walk
Description: The Borg Dyspnea Score is a 10-point scale rating the maximum level of dyspnea experienced after the Six-Minute Walk Test. Scores range from 0 (for the best condition) to 10 (for the worst condition).
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 6
units on a scale | 0.67 (0.52)
Statistical Analysis 1: Comparison: Treprostinil Sodium; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.13, Wilcoxon signed-rank test

4. Secondary Outcome: Change in Score on Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR)
Description: The Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR), a validated PAH-specific instrument consisting of 65 items used to assess symptoms, functioning and quality of life. The questionnaire is divided into three sections; Symptoms (Scores 0-25; high scores indicate more symptoms), Activity (Score 0-30; low score indicates good functioning)and Quality of Life (0-25; high scores indicate poor QoL). The sum of these scores equates to the Total score (0-80). In the CAMPHOR scores, lower scores indicate improvements.
Time Frame: Baseline and Week 8
Population: Two subjects with a Week 8 visit outside of the visit window are included in the summary. One subject died prior to completing the Week 8 visit. One subject had an incomplete Baseline questionnaire and the CAMPHOR Activity component could not be calculated, therefore N=5 Activity and Total Score Components, and N=6 for Symptom and Quality of Life.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 6
units on a scale
  Symptom Score | -2.5 (2.0)
  Activitity Score | -0.8 (2.6)
  Quality of Life Score | -4.4 (6.7)
  Total Score | -8.0 (8.9)
Statistical Analysis 1: Comparison: Treprostinil Sodium; Changes in mean CAMPHOR scores between Baseline and Week 8 were assessed using the Wilcoxon signed rank test. A two-sided p value of < 0.05 was considered statistically significant. No imputation was used for missing values; Test type: Superiority or Other; p = 0.03, Wilcoxon signed rank test — p value for Symptom Score
Statistical Analysis 2: Comparison: Treprostinil Sodium; Activity Score N=5; Baseline component score could not be calculated for one subject. Changes between Baseline and Week 8 were assessed using the Wilcoxon signed rank test. A two-sided p value of < 0.05 was considered statistically significant. No imputation was used for missing values; Test type: Superiority or Other; p = 1.00, Wilcoxon signed rank test — p value for Activity Score
Statistical Analysis 3: Comparison: Treprostinil Sodium; Quality of Life Score. Changes between Baseline and Week 8 were assessed using the Wilcoxon signed rank test. A two-sided p value of < 0.05 was considered statistically significant. No imputation was used for missing values; Test type: Superiority or Other; p = 0.31, Wilcoxon signed-rank test
Statistical Analysis 4: Comparison: Treprostinil Sodium; Total Score N=5; Baseline Activity component score could not be calculated for one subject. Total Score could not be calculated for this subject. Wilcoxon signed rank test was used to compare the values at Baseline to values at Week 8. A two-sided p value of < 0.05 was considered statistically significant. No imputation was used for missing values; Test type: Superiority or Other; p = 0.13, Wilcoxon signed-rank test

5. Secondary Outcome: Change in Score on Treatment Satisfaction Questionnaire for Medication
Description: The Treatment Satisfaction Questionnaire for Medication (TSQM), a validated generic measure of treatment satisfaction consisting of 14 Likert-response items comprising four domains: Effectiveness, Side Effects, Convenience, and Global Satisfaction. The TSQM was completed at baseline and at Week 8. The TSQM consists of 13 items that made up three specific scales (Effectiveness, Side effects, Convenience) and one global satisfaction scale. TSQM items are scaled using either a 5-point or 7-point scale. Five-point scales are used for unidimensional continua (e.g. extremely satisfied to not at all), while 7-point scales are used for bipolar continua(e.g., extremely positive to extremely negative. Non-neutral midpoints are used for 7-point scales, resulting in a greater range of positive response options than negative options for these items. Scale scores are transformed into scores ranging from 0 to 100, with a higher score indicating more satisfaction.
Time Frame: Baseline and Week 8
Population: Two subjects had a Week 8 visit that was outside of the visit window and are included in the summary. One subject died prior to completing the Week 8 visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 6
units on a scale
  Effectiveness Score | -9.3 (13.0)
  Side-Effects Score | 19.8 (28.9)
  Convenience Score | 22.2 (12.2)
  Global Satisfaction Score | -1.2 (21.4)
Statistical Analysis 1: Comparison: Treprostinil Sodium; Effectiveness Score Changes between Baseline and Week 8 were assessed using the Wilcoxon signed rank test. A two-sided p value of < 0.05 was considered statistically significant. No imputation was used for missing values; Test type: Superiority or Other; p = 0.19, Wilcoxon signed-rank test
Statistical Analysis 2: Comparison: Treprostinil Sodium; Side-Effects Score. Changes between Baseline and Week 8 were assessed using the Wilcoxon signed rank test. A two-sided p value of < 0.05 was considered statistically significant. No imputation was used for missing values; Test type: Superiority or Other; p = 0.19, Wilcoxon signed-rank test
Statistical Analysis 3: Comparison: Treprostinil Sodium; Convenience Score. Changes between Baseline and Week 8 were assessed using the Wilcoxon signed rank test. A two-sided p value of < 0.05 was considered statistically significant. No imputation was used for missing values; Test type: Superiority or Other; p = 0.03, Wilcoxon signed-rank test
Statistical Analysis 4: Comparison: Treprostinil Sodium; Global Satisfaction Score. Changes between Baseline and Week 8 were assessed using the Wilcoxon signed rank test. A two-sided p value of < 0.05 was considered statistically significant. No imputation was used for missing values; Test type: Superiority or Other; p = 0.88, Wilcoxon signed-rank test

6. Secondary Outcome: Change in Total Weekly Time Spent With the Specific Activities Associated With Intravenous Remodulin Therapy Compared to Same Activities With Intravenous Epoprostenol
Description: A Drug Administration Activities Diary, used by subjects to record in detail the amount of time (in minutes) spent on specifically-defined drug preparation/administration activities (e.g. diluting drug, preparing reservoir, and changing tubing), was completed over a 7-day period during the Screening period while on epoprostenol and repeated at Week 7 following transition to Remodulin. Drug Administration Activities Diary results are reported as average time per week spent on drug administration activities
Time Frame: Baseline and Week 8
Population: Two subjects did not have Week 8 Drug Administration Activity Diaries completed.
  Connect Drug and Total Time Components: N=4; One subject did not have data recorded for Connect drug activities. Total time could not be calculated for this subject.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 5
minutes
  Gather/Set-up | -2.6 (4.0)
  Prepare Drug | -39.4 (12.8)
  Connect Drug | -5.0 (11.3)
  Change Dressing | 0.0 (10.6)
  Total Time | -44.0 (25.2)
Statistical Analysis 1: Comparison: Treprostinil Sodium; Gather/Set-up. Changes between Baseline and Week 8 were assessed using the Wilcoxon signed rank test. A two-sided p value of < 0.05 was considered statistically significant. No imputation was used for missing values; Test type: Superiority or Other; p = 0.25, Wilcoxon signed-rank test
Statistical Analysis 2: Comparison: Treprostinil Sodium; Prepare Drug. Changes between Baseline and Week 8 were assessed using the Wilcoxon signed rank test. A two-sided p value of < 0.05 was considered statistically significant. No imputation was used for missing values; Test type: Superiority or Other; p = 0.06, Wilcoxon signed-rank test
Statistical Analysis 3: Comparison: Treprostinil Sodium; Connect Drug. Changes between Baseline and Week 8 were assessed using the Wilcoxon signed rank test. A two-sided p value of < 0.05 was considered statistically significant. No imputation was used for missing values; Test type: Superiority or Other; p = 0.63, Wilcoxon signed-rank test
Statistical Analysis 4: Comparison: Treprostinil Sodium; Change Dressing. Changes between Baseline and Week 8 were assessed using the Wilcoxon signed rank test. A two-sided p value of < 0.05 was considered statistically significant. No imputation was used for missing values; Test type: Superiority or Other; p = 0.88, Wilcoxon signed-rank test
Statistical Analysis 5: Comparison: Treprostinil Sodium; Total Time. Changes between Baseline and Week 8 were assessed using the Wilcoxon signed rank test. A two-sided p value of < 0.05 was considered statistically significant. No imputation was used for missing values; Test type: Superiority or Other; p = 0.13, Wilcoxon signed-rank test

7. Secondary Outcome: Change in PAH Signs and Symptoms- Fatigue
Description: The presence or absence of fatigue was documented. If present, the intensity of fatigue was rated mild, moderate, or severe.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 6
participants
  Improved | 0
  No Change | 4
  Worsened | 2
Statistical Analysis 1: Comparison: Treprostinil Sodium; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5, Wilcoxon signed-rank test

8. Secondary Outcome: Change From in Signs and Symptoms of PAH- Edema
Description: The presence or absence of edema was documented. If present, the intensity of edema was rated mild, moderate, or severe.
Time Frame: Baseline and Week 8
Measure: Number; unit: participants
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 6
participants
  Improved | 0
  No Change | 3
  Worsened | 3
Statistical Analysis 1: Comparison: Treprostinil Sodium; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.25, Wilcoxon sign-rank test

9. Secondary Outcome: Change in Signs and Symptoms of PAH- Dyspnea
Description: The presence or absence of dyspnea was documented. If present, the intensity of dyspnea was rated mild, moderate, or severe.
Time Frame: Baseline and Week 8
Measure: Number; unit: participants
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 6
participants
  Improved | 1
  No Change | 3
  Worsened | 2
Statistical Analysis 1: Comparison: Treprostinil Sodium; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 1.00, Wilcoxon signed-rank test

10. Secondary Outcome: Change in Signs and Symptoms of PAH- Orthopnea
Description: The presence or absence of orthopnea was documented. If present, the intensity of orthopnea was rated mild, moderate, or severe.
Time Frame: Baseline and Week 8
Measure: Number; unit: participants
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 6
participants
  Improved | 0
  No Change | 4
  Worsened | 2
Statistical Analysis 1: Comparison: Treprostinil Sodium; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.50, Wilcoxon signed-rank test

11. Secondary Outcome: Change in Signs and Symptoms of PAH- Dizziness
Description: The presence or absence of dizziness was documented. If present, the intensity of dizziness was rated mild, moderate, or severe.
Time Frame: Baseline and Week 8
Measure: Number; unit: participants
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 6
participants
  Improved | 0
  No Change | 5
  Worsened | 1
Statistical Analysis 1: Comparison: Treprostinil Sodium; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 1.00, Wilcoxon signed-rank test

12. Secondary Outcome: Change in Signs and Symptoms of PAH- Syncope
Description: The presence or absence of syncope was documented. If present, the intensity of syncope was rated mild, moderate, or severe.
Time Frame: Baseline and Week 8
Measure: Number; unit: participants
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 6
participants
  Improved | 0
  No Change | 6
  Worsened | 0
Statistical Analysis 1: Comparison: Treprostinil Sodium; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 1.00, Wilcoxon signed-rank test

13. Secondary Outcome: Change in Signs and Symptoms of PAH- Chest Pain
Description: The presence or absence of chest pain was documented. If present, the intensity of chest pain was rated mild, moderate, or severe.
Time Frame: Baseline and Week 8
Measure: Number; unit: participants
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 6
participants
  Improved | 0
  No Change | 5
  Worsened | 1
Statistical Analysis 1: Comparison: Treprostinil Sodium; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 1.00, Wilcoxon signed-rank test

14. Secondary Outcome: Patient Impression of Change Questionnaire
Description: A Patient Global Impression of Change Questionnaire, which consists of three items that ask the subject to rate changes (much better, somewhat better, about the same, somewhat worse, much worse) in their symptoms of PAH, the amount of time spent on activities associated with preparing and administering PAH therapy, and their satisfaction with their PAH therapy since transitioning from epoprostenol to intravenous Remodulin was conducted at Week 8 only and responses are reported as frequency distributions.
Time Frame: Week 8
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 6
participants
  Symptoms- Much Better | 0
  Symptoms-Somewhat Better | 2
  Symptoms- About the Same | 3
  Symptoms- Somewhat Worse | 1
  Symptoms-Much Worse | 0
  Time Spent- Much Less | 3
  Time Spent- Somewhat Less | 3
  Time Spent- About the Same | 0
  Time Spent- Somewhat More | 0
  Time Spent- Much More | 0
  Satisfaction- Much More Satisfied | 1
  Satisfaction- More Satisfied | 3
  Satisfaction- About the Same | 1
  Satisfaction- Less Satisfied | 1
  Satisfaction- Much Less Satisfied | 0

ADVERSE EVENTS:
Time Frame: Adverse events were assessed upon initiation of Remodulin through to the end of study (Week 8)
Description: Since subjects were transitioning from an existing prostacyclin therapy, prostacylin-class side effects ongoing at Baseline prior to transition were recorded separately on the specific Prostacyclin Side Effects Questionnaire. Events which increased in severity from Baseline were captured and reported as AEs.
Arm/Group | Treprostinil Sodium
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treprostinil Sodium (N=7)
Abdominal pain (Gastrointestinal disorders) | 1 (1) — Subject was hospitalized for abdominal pain, nausea, vomiting and dehydration and subsequently died. The investigator assessed the relationship to the study drug as not reasonably attributable to the study drug.
Bacteraemia (Infections and infestations) | 1 (1) — One subject was hospitalized for bacteraemia attributed to Remodulin.
Dehydration (Metabolism and nutrition disorders) | 1 (1) — Subject was hospitalized for abdominal pain, nausea, vomiting and dehydration and subsequently died. The investigator assessed the relationship to the study drug as not reasonably attributable to the study drug.
Nausea (Gastrointestinal disorders) | 1 (1) — Subject was hospitalized for abdominal pain, nausea, vomiting and dehydration and subsequently died. The investigator assessed the relationship to the study drug as not reasonably attributable to the study drug.
Vomiting (Gastrointestinal disorders) | 1 (1) — Subject was hospitalized for abdominal pain, nausea, vomiting and dehydration and subsequently died. The investigator assessed the relationship to the study drug as not reasonably attributable to the study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treprostinil Sodium (N=7)
Headache (Nervous system disorders) | 5 (6)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (4)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Infusion site reaction (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The main limitations of this study are the small sample size, open-label design and relatively short duration of follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the Principal Investigator's rights to discuss or publish trial results after the trial is completed.

Any publication of the results of this trial must be consistent with the United Therapeutics publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the Investigator contract.